CLINICAL TRIAL: NCT01601977
Title: Validation of the AVAPS AE Algorithm in Chronic Obstructive Pulmonary Disease: A Non-randomised Pilot Study
Brief Title: Validation of the AVAPS AE Algorithm in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: AVAPS-AE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Patrick Murphy (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor-Investigator, Patrick Murphy, Clinical Research Fellow, Guy's and St Thomas' NHS Foundation Trust
Organization: Guy's and St Thomas' NHS Foundation Trust (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVAPS AE in COPD; NCT01611870 (obsolete NCT alias)
Record Dates: First submitted 2012-05-17; First posted 2012-05-18 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: COPD; OSA
Keywords: COPD; Respiratory failure; NIV; OSA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): AVAPS-AE
  Interventions: Device: AVAPS-AE
- Usual care (Active Comparator): Non-invasive ventilation
  Interventions: Device: Usual care

INTERVENTIONS:
Device: AVAPS-AE — Novel ventilation mode (Omnilab - AVAPS AE algorithm)
  Arms: Intervention
Device: Usual care — Non-invasive ventilation with standard ventilator
  Arms: Usual care

SUMMARY:
COPD continues to be a cause of major morbidity for patients. Those patients who also have respiratory failure and obstructive sleep apnoea are at higher risk of exacerbations and death and have worse health related quality of life than similar COPD patients without respiratory failure.

Treatment options in this group of patients have been limited and data to support the use of machines to assist breathing (non-invasive ventilators) in stable patients are limited. A major limitation of these devices has been patient acceptance and achieving sufficient control of sleep breathing disturbance.

Currently devices are set at a fixed pressure to support the breathing throughout the night. The new software within the trial device will aim to better match the support provided by the machine to that needed by the patient. It is hoped that this may offer enhanced comfort as well as superior control of respiratory failure.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of morbidity and mortality worldwide.

Treatment options for COPD patients consist of medications, such as bronchodilators and anti-inflammatory drugs, pulmonary rehabilitation, long term oxygen therapy (LTOT), lung volume reduction surgery and lung transplantation. Studies have shown that bronchodilators and anti-inflammatory drugs show minor or no benefit on long term outcomes but rather are used mainly for symptomatic relief.1 Pulmonary rehabilitation has been demonstrated to improve functional status and symptoms but there is lacking evidence on long term outcomes of this therapy. 2 Lung volume reduction surgery and lung transplantation is only appropriate for a small number of patients; therefore, there is no demonstration of improved long-term survival rate.3, 4

Of these available therapies, few have been shown to significantly improve long term patient outcomes. For the severe COPD patient, LTOT is the only treatment that demonstrated prolonged survival in controlled studies. 5, 6 But, despite the effectiveness of LTOT, COPD is still characterized by a high morbidity and mortality rate.

Although the treatment of OSA with CPAP therapy has been associated with reduced hospital admissions and exacerbations there are possible adverse consequences on pulmonary mechanics due to exacerbating hyperinflation.

Noninvasive positive pressure ventilation (NPPV) is one therapy that may prove beneficial to stable COPD patients. NPPV is the use of positive pressure ventilation administered via a nasal or full face mask (that covers both the nose and mouth). This type of ventilation has become a well established and increasingly used therapeutic option for patients with hypercapnic respiratory failure (HRF) due to COPD.7

NPPV, used nocturnally, may improve nighttime hypoventilation that is common with COPD patients. An improvement in nocturnal hypoventilation would reset the respiratory center sensitivity for CO2.8 9 This would result in an improvement in daytime gas exchange and sleep quality. It is also known that hyperinflation in patients with COPD increases their work of breathing, thus fatiguing the respiratory muscles.10 It has been suggested that by applying nocturnal NPPV it would allow the respiratory muscles to rest, resulting in muscle function recovery, increased muscle strength, reduced tendency for fatigue and improvement in pulmonary function and gas exchange.11

AVAPS AE AVAPS AE is a mode of therapy (Philips Respironics Inc, Monroeville, PA, USA) with potential advantages over the currently established modes of noninvasive positive pressure ventilation (CPAP and bilevel therapy). This mode of therapy incorporates AVAPS (automated adjustable IPAP setting to maintain target ventilation with a settable rate of change), AutoEPAP and Auto Back up Rate. In particular the automated EPAP algorithm will ensure optimal upper airway patency without exacerbating hyperinflation.

In this study, we are evaluating the AVAPS AE mode as compared to the participant's current mode of ventilation. We believe that these automated parameters will allow better nocturnal ventilatory control to offset the differing elastic and resistive loads imposed by changes in body position during sleep. Furthermore, AVAPS AE will counter the changing ventilatory requirements due to alterations in lung volumes and airway resistance during different stages of sleep. In summary, the AVAPS AE mode will enable automatic adjustment in response to ventilatory changes throughout the night.

Study Objective The objective of this study is to validate the performance of the AVAPS AE therapy in COPD-OSA overlap patients during nocturnal ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Diagnosis of COPD
* Currently using Bilevel device for COPD-OSA overlap syndrome
* Ability to provide consent
* Documentation of medical stability by PI

Exclusion Criteria:

* Subjects, who are acutely ill, medically complicated or who are medically unstable.
* Subjects in whom PAP therapy is otherwise medically contraindicated.
* Subjects who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days.
* Subjects with untreated, non-OSA sleep disorders, including but not limited to; insomnia, periodic limb movement syndrome, or restless legs syndrome (PLMI > 10).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, Principal Investigator — GSTT
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients approached in ventilation clinic and assessed for trial participation. Patients were recruited and scheduled for trial initiation. Once 10 patients completed the study protocol the remaining recruited patients did not start the assessment period.
Groups:
- All Study Participants: Initial study period in usual care then switched to novel ventilation with AVAPS-AE algorithm
Period: Overall Study
Arm/Group | All Study Participants
Started | 10 (5 patients consented for study participation but did not attend for study assessments.)
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study participants had a pre-existing diagnosis of COPD-OSA and were established on NIV for at least 6 months prior to study enrollement. Patients needed to be clinically stable prior to trial initiation.
Groups:
- All Participants: Single arm crossover nonrandomised study
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Control of Nocturnal Hypoventilation
Description: transcutaneous CO2 recording from overnight sleep study whilst using the device at 6 weeks compared to baseline control when using usual device
Time Frame: baseline, 6 week assessment
Measure: Mean (Standard Deviation); unit: kPa
Groups:
- Intervention: Single arm, open labelled study
  Omnilab - AVAPS AE algorithm: Nocturnal NIV via Omnilab device using the AVAPS AE algorithm
- Usual Care: Usual care including non-invasive ventilation
  Usual care: usual care
  crossover trial, as per intervention
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 10 | 10
kPa | 6.5 (1.6) | 6.7 (1.4)

2. Secondary Outcome: Health Related Quality of Life
Description: Severe Respiratory Insufficiency (SRI) questionnaire. Higher scores indicate better quality of life (minimum 0, maximum 100)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 10 | 10
units on a scale | 60 (15) | 59 (16)

3. Secondary Outcome: Health Related Quality of Life
Description: as for outcome 2
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 10 | 10
units on a scale | 61 (17) | 59 (16)

4. Secondary Outcome: Total Sleep Time
Description: Full polysomnography performed at baseline (usual device) and 6 weeks (trial device) to examine TST
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 10 | 10
minutes | 330 (72) | 306 (72)

5. Secondary Outcome: Control of Nocturnal Hypoventilation
Description: mean tcCO2
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 10 | 10
kPa | 6.4 (1.7) | 6.5 (1.4)

6. Secondary Outcome: Exercise Capacity
Description: 6 minute walk test
Time Frame: 6 weeks
Population: 1 patient declined to complete the walking test
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 9 | 9
m | 190 (63) | 175 (72)

7. Secondary Outcome: Exacerbation Frequency
Description: patient reported exacerbations following 6 weeks of device usage
Time Frame: 6 weeks
Measure: Number; unit: exacerbations
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 10 | 10
exacerbations | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during device usage.
Description: All patients under went clinical review to obtain adverse event data at study assessments
Groups:
- Usual Care: Usual care including non-invasive ventilation
  Usual care: usual care
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Non-randomised controlled study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes